CLINICAL TRIAL: NCT03978403
Title: A Randomized Open-label Four-way Crossover Study of Pharmacokinetics, Safety, and Tolerability of 3 Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes With Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers
Brief Title: A Four-way Crossover Study of 3 Formulations of M207 With Intranasal Zolmitriptan in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zosano Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP-2019-002
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Migraine
Keywords: Pharmacokinetics; Healthy; Volunteer
MeSH Terms: conditions — Migraine Disorders | interventions — zolmitriptan; Nasal Sprays

STUDY DESIGN:
Intervention Model Description: Subjects are randomized to receive one of four treatment sequences of four open-label treatments 48 hours apart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ABDC (Experimental): A: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "Sled" coater packaged in foil pouches; B: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "MACAP" coater packaged in foil cups; C: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "miniMac" coater packaged in foil cups; D: Zolmitriptan nasal 2.5 mg/0.1 mL single dose
  Interventions: Drug: M207 3.8 mg "Sled" (two 1.9 mg patches made on a "Sled" coater, foil pouches); Drug: M207 3.8 mg "MACAP" (two 1.9 mg patches made on a "MACAP" coater, foil cups); Drug: M207 3.8 mg "MiniMac" (two 1.9 mg patches made on a "MiniMac" coater, foil cups; Drug: Zolmitriptan 2.5 mg/0.1 mL nasal spray [ZOMIG] single dose
- BCAD (Experimental): A: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "Sled" coater packaged in foil pouches; B: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "MACAP" coater packaged in foil cups; C: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "miniMac" coater packaged in foil cups; D: Zolmitriptan nasal 2.5 mg/0.1 mL single dose
  Interventions: Drug: M207 3.8 mg "Sled" (two 1.9 mg patches made on a "Sled" coater, foil pouches); Drug: M207 3.8 mg "MACAP" (two 1.9 mg patches made on a "MACAP" coater, foil cups); Drug: M207 3.8 mg "MiniMac" (two 1.9 mg patches made on a "MiniMac" coater, foil cups; Drug: Zolmitriptan 2.5 mg/0.1 mL nasal spray [ZOMIG] single dose
- CDBA (Experimental): A: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "Sled" coater packaged in foil pouches; B: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "MACAP" coater packaged in foil cups; C: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "miniMac" coater packaged in foil cups; D: Zolmitriptan nasal 2.5 mg/0.1 mL single dose
  Interventions: Drug: M207 3.8 mg "Sled" (two 1.9 mg patches made on a "Sled" coater, foil pouches); Drug: M207 3.8 mg "MACAP" (two 1.9 mg patches made on a "MACAP" coater, foil cups); Drug: M207 3.8 mg "MiniMac" (two 1.9 mg patches made on a "MiniMac" coater, foil cups; Drug: Zolmitriptan 2.5 mg/0.1 mL nasal spray [ZOMIG] single dose
- DACB (Experimental): A: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "Sled" coater packaged in foil pouches; B: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "MACAP" coater packaged in foil cups; C: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "miniMac" coater packaged in foil cups; D: Zolmitriptan nasal 2.5 mg/0.1 mL single dose
  Interventions: Drug: M207 3.8 mg "Sled" (two 1.9 mg patches made on a "Sled" coater, foil pouches); Drug: M207 3.8 mg "MACAP" (two 1.9 mg patches made on a "MACAP" coater, foil cups); Drug: M207 3.8 mg "MiniMac" (two 1.9 mg patches made on a "MiniMac" coater, foil cups; Drug: Zolmitriptan 2.5 mg/0.1 mL nasal spray [ZOMIG] single dose

INTERVENTIONS:
Drug: M207 3.8 mg "Sled" (two 1.9 mg patches made on a "Sled" coater, foil pouches) — M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min wear time made on a "Sled" coater and packaged in foil pouches
  Other Names: Treatment A
Drug: M207 3.8 mg "MACAP" (two 1.9 mg patches made on a "MACAP" coater, foil cups) — M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min wear time made on a "MACAP" coater and packaged in foil cups
  Other Names: Treatment B
Drug: M207 3.8 mg "MiniMac" (two 1.9 mg patches made on a "MiniMac" coater, foil cups — M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min wear time made on a "miniMac" coater and packaged in foil pouches
  Other Names: Treatment C
Drug: Zolmitriptan 2.5 mg/0.1 mL nasal spray [ZOMIG] single dose — Zolmitriptan 2.5 mg/0.1 mL nasal spray [ZOMIG] single dose
  Other Names: Treatment D; Zomig Nasal Spray

SUMMARY:
This is a single-center, open-label, randomized, four-way crossover study. Subjects will receive the four study treatments once, followed by in-clinic monitoring and extensive pharmacokinetic analysis. Dosing occurs ~48 hours apart from patch application, in randomized order. Subjects will have final assessment and be dismissed from the study.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, four-way crossover study. Each subject will receive each of the four study treatments once, followed by in-clinic monitoring and extensive blood sample collection for pharmacokinetic analysis.

Dosing will occur approximately 48 hours apart from the time of patch application, until completion of dosing in randomized order per the treatment sequence schedule. Plasma samples from the dosing days will be sent to the analytical laboratory for analysis and tolerability for each of the dose levels will be summarized.

After completion of the four dosing days, subjects will be assessed one final time and dismissed from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men 18 to 50 years of age (inclusive)
2. Good general health with no clinically significant abnormalities as determined by medical history, physical examination, complete blood count, blood chemistry, urinalysis, and ECG.
3. Negative urine drug and alcohol screens and negative serum pregnancy tests (for female subjects) at screening and admission/baseline visit.
4. Consent of female subjects to use a medically effective method of contraception throughout the entire study period and for 30 days after the subject completes the study. Medically effective methods of contraception that may be used by the subject include abstinence, use of diaphragm and spermicide, intrauterine device (IUD), rings, condom and vaginal spermicide, hormonal contraceptives (subjects must be stable on hormonal contraceptives for at least 3 months prior to screening), surgical sterilization (hysterectomy, bilateral tubal ligation, hysteroscopic sterilization) and post-menopausal (≥ 2 years of amenorrhea).
5. Ability to read, understand, and provide written informed consent that they understand the purpose of the study and procedures required for the study before enrolling in the study, and willingness to comply with all study procedures and restrictions.

Exclusion Criteria:

1. Evidence of significant history of hepatic, reproductive, gastrointestinal, renal, bleeding, or hematological disorders including coagulation, pulmonary, neurological, respiratory, endocrine, or cardiovascular system abnormalities (especially hypertension, peripheral vascular disease, coronary artery disease, transient ischemic attacks, or cardiac rhythm abnormalities), psychiatric disorders, acute infection, or other conditions that would interfere with study participation or with the absorption, distribution, metabolism, or excretion of drugs.
2. Presence of three or more of the following CAD risk factors for cardiovascular disease:

   A. Current tobacco use (subjects who have smoked within 30 days of screening)

   B. Hypertension (systolic BP > 140 or diastolic BP > 90) or receiving anti-hypertensive medication for treatment of hypertension

   C. Hyperlipidemia - LDL > 159 mg/dL and/or HDL < 40 mg/dL (or on prescribed anti-cholesterol treatment)

   D. Family history of premature coronary artery disease (CAD) (< 55 years of age in male first-degree relatives or < 65 years of age in female first degree relatives)

   E. Diabetes mellitus
3. Any contraindication to zolmitriptan administration including:

   * History of coronary artery disease or coronary vasospasm
   * Symptomatic Wolf-Parkinson-White syndrome or other cardiac accessory conduction pathway disorders
   * History of stroke, transient ischemic attack, or hemiplegic or basilar migraine
   * Peripheral Vascular Disease
   * Ischemic bowel disease
   * Hypertension (greater than or equal to 140/90 mmHg at either the screening or admission/baseline visit
   * Any history of hepatic impairment defined as alanine transaminase > 150 U/L, aspartate aminotransferase > 130 U/L or bilirubin > 2 times the upper limit of normal
4. History of contact dermatitis or known dermatological disorders that would interfere with the study procedures or assessments
5. Planned participation in activities which cause inflammation, irritation, sunburn, lesions, or tattoos at the intended application sites from 2 weeks prior to dosing through their last day of study participation
6. Use of any prescription anticoagulant within 1 month prior to the first dose
7. Use of prescription and over the counter medications within one week of dosing other than the following:

   * Hormone Replacement Therapy (HRT)
   * Birth control pills, patches, IUD, rings, injections, or implants (all hormonal contraceptives) are allowed provided the dose has been stable for at least three months prior to screening and may be continued throughout the study
   * Proton Pump Inhibitors (PPIs)
   * Antihistamines
   * Intermittently used NSAIDS
   * Acetaminophen if medically necessary (not more than 1000 mg/day)
   * Exceptions may be allowed on a case by case basis
8. Subject has a known allergy or sensitivity to zolmitriptan or its derivatives or formulations
9. Subject has a known allergy or sensitivity to tapes or adhesives
10. Use of any other investigational compound within 30 days of planned study drug dosing
11. Current use or history of drug and/or alcohol abuse within 6 months of screening and deemed to be clinically significant by the investigator
12. History of nasal pathology (e.g., polyps) or abnormal nasal exam deemed to be clinically significant by the investigator
13. Body Mass Index (BMI) lower than 18 kg/m2 or greater than 35 kg/m2
14. If, in the opinion of the investigator, the subject is not suitable for the study
15. Any positive urine drug screen result or alcohol test
16. Subject currently smokes or is a nicotine a user

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Kellerman, PharmD, Study Director — Zosano Pharma Corporation
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ABDC; BCAD; CDBA; DACB: A: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "Sled" coater and packaged in foil pouches; B: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "MACAP" coater and packaged in foil cups; C: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "miniMac" coater and packaged in foil cups; D: Zolmitriptan nasal 2.5 mg/0.1 mL single dose
Period: Overall Study
Arm/Group | ABDC | BCAD | CDBA | DACB
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABDC | BCAD | CDBA | DACB | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (9.69) | 42.2 (4.36) | 35.3 (10.09) | 39.5 (9.87) | 38.7 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 12
  Male | 3 | 3 | 3 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 4 | 4 | 19
  Not Hispanic or Latino | 1 | 0 | 2 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 5 | 6 | 6 | 5 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 24
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 27.153 (3.9165) | 27.118 (3.1446) | 26.523 (4.8929) | 27.242 (2.6340) | 27.009 (3.5044)

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: maximum observed plasma concentration
Time Frame: pre-dose, 2, 5, 10, 15, 20, 30, 45, 60, 90 minutes; 2, 4 , 8, 12, and 24 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Groups:
- M207 3.8 mg (Sled): A: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "Sled" coater and packaged in foil pouches
- M207 3.8 mg (MACAP): B: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "MACAP" coater and packaged in foil cups
- M207 3.8 mg (MiniMac): C: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "miniMac" coater and packaged in foil cups
- Zolmitriptan 2.5 mg (Intranasal): D: Zolmitriptan intranasal 2.5 mg/0.1 mL single dose
Arm/Group | M207 3.8 mg (Sled) | M207 3.8 mg (MACAP) | M207 3.8 mg (MiniMac) | Zolmitriptan 2.5 mg (Intranasal)
Number analyzed (Participants) | 24 | 24 | 24 | 24
pg/mL | 11670 (30.7) | 9861 (93.6) | 11680 (66.3) | 3705 (43.0)

2. Primary Outcome: Adverse Events
Description: Subjects with treatment emergent adverse events
Time Frame: 48 hours
Population: Subjects who received treatment
Measure: Count of Participants; unit: Participants
Groups:
- M207 e.8 mg (MiniMac): C: M207 3.8 mg administered as two 1.9 mg upper arm patches 30 min made on a "miniMac" coater and packaged in foil cups
Arm/Group | M207 3.8 mg (Sled) | M207 3.8 mg (MACAP) | M207 e.8 mg (MiniMac) | Zolmitriptan 2.5 mg (Intranasal)
Number analyzed (Participants) | 24 | 24 | 24 | 24
Participants | 18 | 15 | 13 | 4

3. Primary Outcome: Tmax
Description: Time to maximum concentration
Time Frame: pre-dose, 2, 5, 10, 15, 20, 30, 45, 60, 90 minutes; 2, 4 , 8, 12, and 24 hours post-dose
Measure: Median (Full Range); unit: hour
Arm/Group | M207 3.8 mg (Sled) | M207 3.8 mg (MACAP) | M207 3.8 mg (MiniMac) | Zolmitriptan 2.5 mg (Intranasal)
Number analyzed (Participants) | 24 | 24 | 24 | 24
hour | 0.529 [0.34 to 0.76] | 0.577 [0.04 to 0.79] | 0.575 [0.33 to 0.77] | 2.000 [0.56 to 4.00]

ADVERSE EVENTS:
Time Frame: 8 days total, 48 hours per intervention
Arm/Group | M207 3.8 mg (Sled) | M207 3.8 mg (MACAP) | M207 3.8 mg (MiniMac) | Zolmitriptan 2.5 mg (Intranasal)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 18/24 | 15/24 | 13/24 | 4/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M207 3.8 mg (Sled) (N=24) | M207 3.8 mg (MACAP) (N=24) | M207 3.8 mg (MiniMac) (N=24) | Zolmitriptan 2.5 mg (Intranasal) (N=24)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0
Abdominal ditension (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Application site discolouration (General disorders) | 12 | 12 | 9 | 0
Application site pain (General disorders) | 1 | 1 | 2 | 0
Feeling hot (General disorders) | 1 | 1 | 0 | 0
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0
Vessel puncture site swelling (General disorders) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal sstiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesea (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT03978403/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT03978403/SAP_001.pdf